CLINICAL TRIAL: NCT05314816
Title: Clinical Impact of a Multiplex PCR Blood Culture Identification Panel in Early Identification of Positive Blood Cultures in Pediatric Patients in Guatemala
Brief Title: Rapid Blood Culture Identification Panel in Pediatric Patients in Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-0464
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Bacteremia; Sepsis
Keywords: bacteremia; sepsis; antimicrobial resistance; BCID2; multiplex PCR; pediatric
MeSH Terms: conditions — Bacteremia; Sepsis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Blood culture identification panel (Experimental): BioFire BCID2 (Blood culture identification panel) will be performed on positive blood culture specimens.
  Interventions: Diagnostic Test: Blood culture identification panel
- Concurrent control (No Intervention): Standard blood culture process will be performed concurrently on select positive blood culture specimens during the study period. BCID2 will NOT be performed on these specimens.
- Retrospective control (No Intervention): Standard blood culture process was performed prior to the study period.

INTERVENTIONS:
Diagnostic Test: Blood culture identification panel — multiplex PCR panel to be performed on positive blood cultures
  Other Names: BCID2; BioFire BCID2 Panel; BioFire FilmArray
  Arms: Blood culture identification panel

SUMMARY:
The purpose of this study is to assess the clinical impact of a rapid multiplex PCR blood culture identification panel on time to optimal antimicrobial therapy when compared to conventional microbiological culture methods in children hospitalized in a low resource setting in Guatemala City.

DETAILED DESCRIPTION:
A retrospective review of positive blood cultures was performed on pediatric patients at a tertiary hospital in Guatemala City. These will serve as retrospective controls. The prospective portion of this study will implement the BioFire FilmArray blood culture identification panel (BCID2). Laboratory technicians will perform BCID2 simultaneously with standard culture after it flags positive on the automated blood culture system. BCID2 will be performed on those blood culture specimens that become positive during normal laboratory daytime working hours. Those specimens that become positive overnight will not have the BCID2 performed and will serve as concurrent controls. Physicians will be notified of panel results for the BCID2 intervention group and standard culture results per current laboratory protocol. This study will compare time to optimal antimicrobial therapy (primary outcome), as well as secondary outcome measures, between the intervention group and the 2 control groups.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years of age
* First positive blood culture during the hospitalization

Exclusion Criteria:

* Non-blood specimens
* Repeat positive blood cultures from the same admission
* Patients who expire prior to positive culture
* Outpatient blood cultures

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 479 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Dominguez, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Hospital Roosevelt, Guatemala City, Guatemala

REFERENCES:
- [Derived] Graff KE, Galvez N, Lamb MM, Cortes R, Sanchez Villeda EA, Calvimontes DM, Melgar MA, Olson D, Asturias EJ, Dominguez SR. Evaluating the Clinical Impact of the BCID2 Panel and Antimicrobial Stewardship in Pediatric Bloodstream Infections: A Pragmatic Trial in Guatemala. Pediatr Infect Dis J. 2025 Nov 1;44(11):1051-1058. doi: 10.1097/INF.0000000000004937. Epub 2025 Aug 1. PMID 40880253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control
Started | 159 | 221 | 99
Analyzed in Concurrent Control Group (enrolled in intervention, but analyzed in concurrent control group because they did not receive the allocated intervention) | 6 | 0 | 0
Completed | 141 | 213 | 98
Not Completed | 18 | 8 | 1
Not completed — Lost to Follow-up | 5 | 0 | 1
Not completed — Protocol Violation | 13 | 8 | 0

BASELINE CHARACTERISTICS:
Population: 452 patients completed the study and were analyzed. Note that 6 patients were originally enrolled in the BCID group, but ultimately analyzed in the concurrent control group as they did not receive the intervention as allocated. These 6 patients crossed over from the BCID group into the concurrent control group for the analysis, leaving 135 in the BCID and 219 in the concurrent control group for the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control | Total
Number analyzed (Participants) | 135 | 219 | 98 | 452
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 135 | 219 | 98 | 452
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 1 [0.3 to 22.1] | 1 [0.3 to 16.4] | 0 [0 to 9] | 0.9 [0.2 to 14.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 99 | 36 | 196
  Male | 74 | 120 | 62 | 256
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Guatemala | 135 | 219 | 98 | 452
Antecedent medical conditions [Count of Participants; unit: Participants]
  No antecedent medical conditions | 70 | 114 | 25 | 209
  One or more medical condition | 65 | 105 | 73 | 243
Central line [Count of Participants; unit: Participants] | 67 | 132 | 70 | 269
ICU stay [Count of Participants; unit: Participants] | 68 | 133 | 73 | 274

OUTCOME MEASURES:

1. Primary Outcome: Time to Optimal Antimicrobial Therapy
Description: Calculated from the time of blood culture draw to the time that optimal antimicrobial therapy is started. Optimal antimicrobial therapy is defined based on pre-determined organism-antimicrobial guidelines.
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control
Number analyzed (Participants) | 135 | 219 | 98
hours | 31.1 [0 to 150] | 117.7 [0 to 248.4] | 90.0 [4.3 to 158.0]

2. Secondary Outcome: Time to Organism Identification
Description: Calculated from the time of blood culture draw to the time of organism identification.
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control
Number analyzed (Participants) | 135 | 219 | 98
hours | 22.6 [20.3 to 28] | 79.8 [61.7 to 104.5] | 76.8 [66.9 to 91.0]

3. Secondary Outcome: Time to Effective Antimicrobial Therapy
Description: Calculated from the time of blood culture draw to the time that the effective therapy is started. Effective therapy is determined based on susceptibilities of the organism.
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control
Number analyzed (Participants) | 135 | 219 | 98
hours | 0 [0 to 33.9] | 0.2 [0 to 120.2] | 3.0 [0 to 89.0]

4. Secondary Outcome: All-cause Mortality
Description: 30 day mortality
Time Frame: 30 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control
Number analyzed (Participants) | 135 | 219 | 98
Participants | 14 | 30 | 18

5. Secondary Outcome: Length of Hospital Stay
Time Frame: 30 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control
Number analyzed (Participants) | 135 | 219 | 98
days | 17 [11 to 30] | 20 [11 to 30] | 17 [10 to 30]

6. Secondary Outcome: Intensive Care Unit Days
Description: Days in the ICU
Time Frame: 30 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control
Number analyzed (Participants) | 135 | 219 | 98
days | 14.3 [7.5 to 26.2] | 14.8 [8.5 to 28.0] | 9.0 [6.0 to 15.5]

ADVERSE EVENTS:
Time Frame: 30 days
Description: 452 patients completed the study and were analyzed. Note that 6 patients were originally enrolled in the BCID group, but ultimately analyzed in the concurrent control group as they did not receive the intervention as allocated. These 6 patients crossed over from the BCID group into the concurrent control group for the analysis, leaving 135 in the BCID and 219 in the concurrent control group for the analysis.
Arm/Group | Blood Culture Identification Panel | Concurrent Control | Retrospective Control
All-Cause Mortality (participants affected / at risk) | 14/135 | 30/219 | 18/98
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/219 | 0/98
Other Adverse Events (participants affected / at risk) | 0/135 | 0/219 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT05314816/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT05314816/SAP_001.pdf